CLINICAL TRIAL: NCT06815315
Title: A Formative, Mixed-Methods Evaluation Assessing the Acceptability, Feasibility, and Effectiveness of Micronutrient Interventions Among Adolescents in Mozambique
Brief Title: Evaluating of the Impact of Micronutrient Interventions Among Adolescents in Mozambique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: World Vision US (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WorldVision; 218961 (Other Grant/Funding Number: World Vision Canada)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Anemia
Keywords: Vitamins; Supplements; Iron; Folic Acid; Mozambique; Micronutrients; Adolescents
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: We conducted a two-arm cluster-randomized trial in three secondary schools, enrolling 28 girls' clubs (14 per arm), with each club consisting of approximately 18 girls aged 13 to 20 years. Using constrained sampling to balance for age and school, clubs were randomly assigned to one of two intervention groups: (1) Multiple Micronutrient Supplementation (MMS) for five months plus a Nutrition Curriculum, or (2) Iron and Folic Acid Supplementation (IFAS) plus a Nutrition Curriculum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multiple Micronutrient Supplementation (MMS) Arm (Active Comparator): The adolescent girls randomly assigned to the MMS arm consumed MMS for four months and participated in girls' clubs where they received nutrition messages.
  Interventions: Dietary Supplement: Multiple micronutrient supplementation; Behavioral: Adolescent Nutrition Curriculum
- Iron Folic Acid Supplementation (IFAS) Arm (Active Comparator): The adolescent girls randomly assigned to the IFAS arm consumed IFAS for four months and participated in girls' clubs where they received nutrition messages
  Interventions: Dietary Supplement: Iron Folic Acid Supplementation; Behavioral: Adolescent Nutrition Curriculum

INTERVENTIONS:
Dietary Supplement: Multiple micronutrient supplementation — The multiple micronutrient supplementation composition follows the United Nations International Multiple Micronutrient Antenatal Preparation. Each MMS tablet contains 15 micronutrients, including iron (30mg), folic acid (400 mcg), Vit A, Retinol (800 RE), vit D (200 IU), vit E (10 mg), vit C (70 mg), vit B1 (1.4 mg), vit B2 (1.4 mg), vit B6 (1.9 mg), vit B12 (2.6 mcg), niacin (18 mg), zinc (15 mg), copper (2 mg), iodine (150 mcg), selenium (65 mcg) and is consumed daily.
  Arms: Multiple Micronutrient Supplementation (MMS) Arm
Dietary Supplement: Iron Folic Acid Supplementation — One IFAS tablet contains Iron (60 mg) and Folic Acid (2800 μg) and is taken weekly.
  Arms: Iron Folic Acid Supplementation (IFAS) Arm
Behavioral: Adolescent Nutrition Curriculum — The Adolescent Nutrition Curriculum includes five modules focused on promoting healthy behaviors to enhance nutrition, with an emphasis on consuming iron-rich foods.

SUMMARY:
This purpose of this study is to assess effects of iron and folic acid supplementation and multiple micronutrient supplementation on anemia status and the impact of a nutrition curriculum on diet diversity and anemia knowledge among adolescent girls.

DETAILED DESCRIPTION:
This study aimed to implement and evaluate micronutrient supplementation interventions to improve adolescent nutrition, health, and education in Mozambique. In conjunction with the Mozambique Ministries of Health, Education and Culture, we conducted a two-arm cluster-randomized trial in three secondary schools, enrolling 28 girls' clubs (14 per arm). Each club was comprised of around 18 girls aged 13 to 20 years. Using constrained sampling to balance for age and school, clubs were randomly assigned to one of two intervention groups: 1) Multiple Micronutrient Supplementation (MMS) for five months plus a Nutrition Curriculum, or 2) Iron and Folic Acid Supplementation (IFAS) plus a Nutrition Curriculum. Girls enrolled in the MMS arm consumed supplements daily for 4 months at home and weekly nutrition messages delivered through the clubs. Girls enrolled in the IFAS arm consumed supplements once a week for 4 months at school (the standard of care) and weekly nutrition messages delivered through the clubs. The study evaluated the effects of MMS and IFAS on anemia status and the impact of the nutrition curriculum on diet diversity and anemia knowledge.

ELIGIBILITY:
Inclusion Criteria:

Adolescents aged 13-20 years Enrolled in secondary school at study initiation Member of an IMPACT+ Girls Club at one of the participating schools Consent provided by the parent Assent provided by the adolescent

Exclusion Criteria:

No informed consent from parent or assent from adolescent Self-reported pregnancy

Ages: 13 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 490 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Anemia Status | 6 months
  Anemia is defined as hemoglobin level <10 g/dL

SECONDARY OUTCOMES:
Anemia Knowledge | 6 months
  Changes in knowledge from baseline to endline around anemia causes and strategies to prevent anemia.
Minimum Dietary Diversity Score | 6 months
  The minimum dietary diversity score measures girls and women who 10 possible food groups over a 24-hour recall period are classified as having minimally adequate diet diversity.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Bauler, DrPH(c), Principal Investigator — World Vision International
Locations (1):
- World Vision Monapo Field Office, Monapo, Nampula, Mozambique

IPD SHARING:
Plan to Share IPD: Undecided
With permission from the Mozambique Ministry of Health Commitee for Bioethics, the quantitative dataset supporting the conclusions of this study can be found in the Humanitarian Data Exchange at https://data.humdata.org.

REFERENCES:
- See also: The paper on photovoice published in the Emergency Nutrition Action Field Exchange describes the methodology and findings we used to develop and refine the Nutrition Curriculum. The Nutrition Curriculum is one of the interventions tested in this CRT. — https://www.ennonline.net/fex/74/photovoice-enhancing-health-and-nutrition-mozambiques